CLINICAL TRIAL: NCT05179551
Title: Proximal Medial Gastrocnemius Recession for Chronic Mid-Portion Achilles Tendinopathy; A Multicenter, Prospective Cohort Study.
Brief Title: Achillestendinopathy Treated With Proximal Medial Gastrocnemius Recession
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK244374
Record Dates: First submitted 2021-10-21; First posted 2022-01-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Achilles Tendinopathy; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proximal Medial Gastrocnemius Recession Surgery (Experimental): Patients will be operated with Proximal Medial Gastrocnemius Recession Surgery (PMGR) ad modum Barouk.
  Interventions: Procedure: Proximal Medial Gastrocnemius Recession

INTERVENTIONS:
Procedure: Proximal Medial Gastrocnemius Recession — . A 3-4 cm transverse skin incision is made in the popliteal fossa, the superficial fascia is opened, and the medial gastrocnemius with its tendon (aponeurosis) is located. The tendon is then cut while lifting it with clamps, and care is taken to cut only the white tendon while sparing the underlying muscle. While performing a dorsiflexion movement of the ankle, careful palpation of the muscle is done to ensure that all tendon strands are cut completely. The incision is closed in layers, and only soft dressings applied
  Other Names: PMGR

SUMMARY:
This is a prospective cohort study that will follow 60 patients treated with Proximal Medial Gastrocnemius Recession for Chronic Mid-Portion Achilles Tendinopathy for 5 years postoperatively.

DETAILED DESCRIPTION:
Mid Portion Achilles Tendinopathy is a condition that usually resolves by itself without any kind of intervention. If the condition becomes chronic, eccentric training guided by a physical therapist seems to be the best non-surgical intervention. Surgical treatment has shown varying results and no gold-standard exists.

Tightness in the gastrocnemius muscle seems to be a contributing factor for many conditions in the foot and ankle region.

Retrospective material suggest that Proximal Medial Gastrocnemius Recession (PMGR) can be an effective treatment for this condition. No prospective material exists.

This study aims at including 60 patients with Chronic Mid-Portion Achilles Tendinopathy (CMPAT) that is non-responsive to eccentric training. Patients will be PMGR-surgery and followed for 5 years with PROMS, muscle function test and MRI scans.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-75 years.
2. Diagnosis CMPAT verified clinically by orthopedic surgeon. Symptoms must include mid-portion pain in the Achilles, swelling and reduced tolerance for weightbearing.
3. Verified diagnosis with MRI findings representing pathologic processes of tendon degeneration and repair (13). MRI no older than 12 months.
4. Duration of symptoms must be at least 12 months.
5. Isolated gastrocnemius tightness must be verified with the Silfverskiölds test before inclusion. The Silfverskiöld test is considered positive if ankle dorsiflexion is restricted to 5 degrees or less with the knee extended, and there is an increase of ankle dorsiflexion of at least 10 degrees when flexing the knee.
6. At least three months of conventional physical therapy with eccentric training must have been tried without providing relief of symptoms.

Exclusion criteria:

1. Previous history of complete Achilles tendon rupture.
2. Other combined pathologies in the Achilles tendon of calf (Sequela from trauma, infections, cancer etc.).
3. Insertional Achilles tendinopathy.
4. Previously undergone surgery in affected tendon.
5. Patients with severe talocrural pathology or serious malalignment of foot and ankle.
6. Severely reduced peripheral circulation.
7. History of alcoholism, drug abuse, psychological or other emotional problems likely to jeopardize informed consent.
8. Patients with a contraindication/non-compliance for MRI examination.
9. History of allergic reaction/anaphylactic reaction to local anesthetics.
10. Not able to read and/or speak a Scandinavian language or English adequately.
11. Other serious comorbidity that makes surgery unadvisable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VISA-A - Victorian Institute of Sport Assessment- Achilles Questionnaire | Baseline
  A PROM validated for patients with achilles tendon disorders
VISA-A - Victorian Institute of Sport Assessment- Achilles Questionnaire | 3 months
  A PROM validated for patients with achilles tendon disorders
VISA-A - Victorian Institute of Sport Assessment- Achilles Questionnaire | 1 year
  A PROM validated for patients with achilles tendon disorders
VISA-A - Victorian Institute of Sport Assessment- Achilles Questionnaire | 2 years
  A PROM validated for patients with achilles tendon disorders
VISA-A - Victorian Institute of Sport Assessment- Achilles Questionnaire | 5 years
  A PROM validated for patients with achilles tendon disorders

SECONDARY OUTCOMES:
Achilles Function Test battery | Baseline, 3 months, 2 years
  The test battery consists of three jump tests, a counter movements jump (CMJ), a drop counter movement jump (drop CMJ) and hopping, and two strength tests, concentric toe-raises, eccentric-concentric toe-raises and toe-raises for endurance. All recorded through the MuscleLab software.
Ankle Dorsiflexion pre and postoperatively | Baseline, 3 months, 2 years
  measured with a validated goniometer that measures the ankle's range of motion- The device has been previously tested and found to be valid, reliable, and responsive in detecting isolated gastrocnemius contractures (IGCs). An electric goniometer, Biometrics SG150 (Units 25-26, Biometrics Ltd, Newport, UK), with an accuracy of ±2 degrees and a repeatability of 1 degree will be used. The device will be calibrated before every new participant. Force applied directly beneath the head of the second metatarsal until the end range of dorsiflexion with a dynamometer.
MRI findings pre inclusion versus after 2 years. | Baseline, 2years
  a. Tendon thickness - Thickest point anterior-posteriorly in the sagittal plane in millimeters. Cm2 at thickest point in the axial plane.
VAS | Baseline, 3 months, 1 year, 2 years, 5 years
  Visual Analogue Scale for pain during use of affected leg in the last 24 hours. 0 is no pain. 10 is worst pain imaginable.
Eq-5D | Baseline, 3 months, 1 year, 2 years, 5 years
  Quality of life is measured by the EuroQol questionnaire (EQ-5D). EQ-5D is a validated generic health-related quality-of-life instrument. It consists of two parts: EQ-5D descriptive part and EQ-5D visual analogue scale. The descriptive part includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five possible answers ("no problems", "some problems", and "major problems"). EQ5D VAS is a visual analogue scale of self-related overall health, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Adverse events | Baseline, 3 months, 1 year, 2 years, 5 years
  Infection, thrombosis, nerve injury etc
MRI findings pre inclusion versus after 2 years. | baseline, 2 years
  Reduction of intratendinous signal - YES/NO
Assessment of treatment success - pain | 2 years
  Likert question: I have pain in the achilles tendon of the leg that was operated two years ago.
  1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - physical activity | 2 years
  Likert question: Achilles pain prevents me from performing physical activites
  1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - daily living | 2 years
  Likert question: Achilles pain prevents me from performing activities of daily living
  1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - calf pain | 2 years
  Likert question: I have pain and/or discomfort in the calf muscle that was operated two years ago
  1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree
Assessment of treatment success - other treatments | 2 years
  I have received other treatments for achilles pain since surgery was preformed two years ago YES/NO
Assessment of treatment success - Patient Acceptable Symptom State | 2 years
  If you were to continue having the same level of achilles symptoms in the coming few months, would you consider that acceptable? YES/NO

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (2):
- Norway (2):
  - Oslo University Hospital, Orthopedic Department Ullevål, Oslo
  - Østfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No